CLINICAL TRIAL: NCT05710302
Title: Investigation of the Diagnostic Accuracy of EHMRG Risk Score in Patients With Acute Heart Failure
Brief Title: Prospective Validation of the Emergency Heart Failure Mortality Risk Grade (EHMRG) Score in Patients With Acute Heart Failure in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berkay Ünlü, MD, Marmara University Pendik Training and Research Hospital
Other Study IDs: 09.2022.742
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Heart Diseases; Acute Heart Failure
Keywords: mortality; emergency department; heart failure; hospitalization; risk assessment; discharge planning
MeSH Terms: conditions — Heart Failure; Heart Diseases; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with acute heart failure in the emergency department: Patients with acute heart failure.
  Interventions: Other: Investigation of the diagnostic accuracy of EHMRG risk score in patients with acute heart failure

INTERVENTIONS:
Other: Investigation of the diagnostic accuracy of EHMRG risk score in patients with acute heart failure — Prospective validation of the EHMRG score in patients with acute heart failure in the emergency department

SUMMARY:
In this prospective validation study, researchers investigates accuracy of EHMRG (Emergency Heart Failure Mortality Risk Grade) score in predicting the 7th and 30th day risk of mortality in patients with acute heart failure who applying to the emergency department.

DETAILED DESCRIPTION:
Heart failure is a serious public health problem in the world due to its high morbidity and mortality rate.Turkish Society of Cardiology conducted a prevalence study. The name of the study is HAPPY. Accordingly, the prevalence of heart failure in people over 35 years of age in Turkey is 2.9%.The prevalence of heart failure in Turkey is higher than in European countries.

The incidence of heart failure cases with no obvious symptoms is 4.9% in Turkey. Patients with a diagnosis of heart failure apply to the emergency department frequently. There are scoring studies around the world for patients' hospitalization and discharge.

EHMRG score created and validated by Douglas S. Lee et al. In our study, the accuracy of EHMRG score will be investigated prospectively in patients diagnosed with acute heart failure in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute heart failure in the emergency department

Exclusion Criteria:

* Dialysis dependent patients
* Pregnant patients
* Patients brought to the emergency department with cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute heart failure in the emergency department.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 7 days
  Death within 7 days after emergency department presentation for acute heart failure.
Mortality | 30 days
  Death within 30 days after emergency department presentation for acute heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Berkay UNLU, MD, Principal Investigator — Marmara University School of Medicine Emergency Department
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study plan, collected data and statistical analyzes will be shared with the researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months
Access Criteria: Ethics Committee Approval

REFERENCES:
- [Result] Lee DS, Lee JS, Schull MJ, Grimshaw JM, Austin PC, Tu JV. Design and rationale for the Acute Congestive Heart Failure Urgent Care Evaluation: The ACUTE Study. Am Heart J. 2016 Nov;181:60-65. doi: 10.1016/j.ahj.2016.07.016. Epub 2016 Aug 7. PMID 27823694
- [Result] van Hattem NE, Beeres SLMA, Mertens BJA, Antoni ML, Atsma DE, Schalij MJ, den Haan MC. Emergency Heart failure Mortality Risk Grade may help to reduce heart failure admissions. Neth Heart J. 2022 Sep;30(9):431-435. doi: 10.1007/s12471-022-01661-3. Epub 2022 Mar 11. PMID 35277803
- [Result] Lee DS, Lee JS, Schull MJ, Borgundvaag B, Edmonds ML, Ivankovic M, McLeod SL, Dreyer JF, Sabbah S, Levy PD, O'Neill T, Chong A, Stukel TA, Austin PC, Tu JV. Prospective Validation of the Emergency Heart Failure Mortality Risk Grade for Acute Heart Failure. Circulation. 2019 Feb 26;139(9):1146-1156. doi: 10.1161/CIRCULATIONAHA.118.035509. PMID 30586748
- [Result] Lee DS, Stitt A, Austin PC, Stukel TA, Schull MJ, Chong A, Newton GE, Lee JS, Tu JV. Prediction of heart failure mortality in emergent care: a cohort study. Ann Intern Med. 2012 Jun 5;156(11):767-75, W-261, W-262. doi: 10.7326/0003-4819-156-11-201206050-00003. PMID 22665814
- See also: Design and rationale for the Acute Congestive Heart Failure Urgent Care Evaluation: The ACUTE Study. — https://pubmed.ncbi.nlm.nih.gov/27823694/
- See also: Emergency Heart failure Mortality Risk Grade may help to reduce heart failure admissions. — https://pubmed.ncbi.nlm.nih.gov/35277803/
- See also: Prospective Validation of the Emergency Heart Failure Mortality Risk Grade for Acute Heart Failure. — https://pubmed.ncbi.nlm.nih.gov/30586748/
- See also: Prediction of heart failure mortality in emergent care: a cohort study. — https://pubmed.ncbi.nlm.nih.gov/22665814/